CLINICAL TRIAL: NCT04011163
Title: Vital Signs-Integrated Patient-Assisted Intravenous Opioid Analgesia for Post Surgical Pain
Acronym: VPIA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHIC-I2I-1812002
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pain; Respiratory Depression
Keywords: Postoperative pain; Respiratory depression; Bradypnoea; Morphine; Infusion pump
MeSH Terms: conditions — Pain; Respiratory Insufficiency; Pain, Postoperative; Hypoventilation | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VPIA analgesia (Experimental): VPIA pump will be connected to patients after surgery for up to three days. The vital signs (oxygen saturation, respiratory rate, heart rate) will be closely monitored when patients are using VPIA pump. Intravenous medication (morphine) will be given intravenously.
  Interventions: Device: VPIA pump; Drug: Morphine

INTERVENTIONS:
Device: VPIA pump — The pump is a specially designed and manufactured infusion syringe pump for intravenous analgesia. It incorporates the VPIA study regimen to meet the specific requirements of the clinical trial. It is intended to be used only for delivering drugs intravenously.
  Other Names: VPIA delivery system
Drug: Morphine — Intravenous medication used is morphine diluted in normal saline to a concentration of 1mg/ml. This is a standard dilution and are routine drugs used as standard of care.
  Other Names: Morphine Sulphate

SUMMARY:
To meet the unmet need of better and safer pain relief for acute pain in the post-operative setting, a Vital-signs-integrated Patient-assisted Intravenous opioid Analgesia ("VPIA") Delivery System, with novel and intelligent software algorithms and specialised hardware was developed. In the previous project, the investigators have shown that this system has the potential to increase the safety and patient satisfaction with intravenous opioid analgesia. However, opportunities to develop more robust vital signs monitoring with the goal of ensuring continual and effective analgesia are identified.

The primary aim of this proposal is to advance the development of technology (through new features and functionality) and perform clinical evaluation of the VPIA system with a larger sample size to show improvements in patient's satisfaction (pain relief) and robustness of system in terms of vital signs integration. Novel technology using adaptive vital signs controller, integrated with an infusion pump and single finger probe vital signs monitor system will be developed with the aim for commercialisation.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study in 150 adult female subjects that undergo major surgery that require postoperative patient controlled morphine analgesia so as to examine the monitoring performance of oxygen desaturation, respiratory depression and patient satisfaction and user feedback.

Patients who are undergoing elective surgery with plan to use postoperative patient controlled analgesia with morphine will receive study information either at pre-operative assessment clinic or upon admission for surgery if they have not attended the pre-operative assessment clinic. They will be screened for eligibility using the inclusion and exclusion criteria. If eligible for recruitment, the patients will be approached by the investigators for recruitment. Upon successful recruitment of the study, patients will be asked to complete two questionnaires and rate their pre-surgical pain on the numerical rating scale in the pre-anaesthetic evaluation clinic. The general anaesthesia technique and type of analgesia administered intra-operatively will be according to standard practice and is at the discretion of the attending anaesthesiologist. After surgery, patients will be reviewed daily (up to 3 days) in the post-operative wards. They will be asked on questionnaire scoring, pain score, and analgesia information and adverse event, if any.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologist (ASA) physical status I-III;
* Age 21-70 years;
* Receiving patient controlled analgesia of morphine for postoperative analgesia.

Exclusion Criteria:

* Allergy to study drug;
* With significant respiratory disease and obstructive sleep apnea;
* Unwilling to place oxygen saturation and respiratory rate monitoring during study period;
* Unable to comprehend the use of patient controlled analgesia;
* Obstetric patients.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females undergoing gynecologic surgery in KKH will be recruited.
Enrollment: 40 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of a clinically significant bradypnoea | Postoperative period (1 - 3 days)
  The number of events of respiratory rate less than 8 per minute throughout the study period (when the patient is connected to the pump)

SECONDARY OUTCOMES:
Postoperative pain score | Postoperative period (1 - 3 days)
  Pain scores (Numeric Rating Scale 0-10) will be asked, with zero being no pain, and 10 being the worst pain possible.
Patient satisfaction | Postoperative period (1 day, after the use of pump)
  Patient will be asked about their satisfaction level on the pump based on ordinal scale (Strongly disagree, disagree, neutral, agree, strongly agree).
Changes in Hospital Anxiety and Depression Scale (HADS) score | Before surgery (1 day) and postoperative period (1-3 days)
  HADS Anxiety and Depression score before and after surgery. HADS is commonly used by doctors to determine the levels of anxiety and depression that a patient is experiencing. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. For each subscore (anxiety/depression), 0-7 = Normal; 8-10 = Borderline abnormal (borderline case); and 11-21 = Abnormal (case).
EQ-5D-3L score | Before surgery (1 day)
  EQ-5D-3L score before surgery. EQ-5D-3L is a standardized instrument for measuring generic health status. It is made up for two components; health state description and evaluation. The health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension ranging from 1-3. From these five dimensions, EQ-5D index is calculated, having a value between 0-1. The evaluation part involves an analogue scale, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " the worst health you can imagine", and hundred corresponds to "the best health you can imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, MBBS, MMED, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maddox RR, Williams CK, Oglesby H, Butler B, Colclasure B. Clinical experience with patient-controlled analgesia using continuous respiratory monitoring and a smart infusion system. Am J Health Syst Pharm. 2006 Jan 15;63(2):157-64. doi: 10.2146/ajhp050194. No abstract available. PMID 16390930